CLINICAL TRIAL: NCT03570333
Title: Identification and Application of Gingival Mesenchymal Stem Cells for Dental Tissue Regeneration.
Brief Title: Progenitor Potential of Mesenchymal Stem Cells in Palatal Tissue Harvested From Molar and Premolar Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maninder Kaur, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300000607; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2018-06-17; First posted 2018-06-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gingival Recession; Lack of Keratinized Gingiva (Disorder)
Keywords: gingival recession; gingival graft; Palate; Gingival mesenchymal stem cells; molar; premolar
MeSH Terms: conditions — Gingival Recession; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progenitor Potential at Molar site (Experimental): Harvested tissue from the back (molar) part of the palate will be used to extract the gingival mesenchymal cells to test their progenitor potential to differentiate into multiple cell lineage.
  Interventions: Diagnostic Test: progenitor potential of Gingival Mesenchymal cells
- Progenitor Potential at Premolar site (Experimental): Harvested tissue from the front (premolar) part of the palate will be used to extract the gingival mesenchymal cells to test their progenitor potential to differentiate into multiple cell lineage.
  Interventions: Diagnostic Test: progenitor potential of Gingival Mesenchymal cells

INTERVENTIONS:
Diagnostic Test: progenitor potential of Gingival Mesenchymal cells — tissues collected from the molar and premolar sites will be sent to the lab for cell culturing. once in the lab, the tissues will be already separated and labeled (molar) and ( premolar) and then treated to extract the cells from them. then, these cells will be tested for their capacity to form different kinds of cells and tissues ( bone, cartilage, fibers for periodontal ligaments). After this test, results will be collected for how many cells were collected from each tissue sample.

SUMMARY:
The primary purpose of this protocol is to isolate, investigate and compare the regenerative and differentiation potential of mesenchymal stem cells (MSC's) in the gingival (gum) tissue harvested from two different locations from the roof of the mouth (palate), that is from the front part(premolar)and back part(molar). MSC's are known for their capacity to form different kinds of hard and soft tissue including bone, fibers for periodontal ligaments, cementum and dentin, thus this study can help in optimizing their clinical application and transplantation approaches in tissue regeneration.

DETAILED DESCRIPTION:
Various types of stem cells, specifically Mesenchymal Stem Cells (MSCs) have been thoroughly investigated for their role in tissue engineering, regenerative medicine and regeneration of the attachment apparatus (bone, cementum, periodontal ligament) of the tooth (that is lost due to periodontal disease) through multidisciplinary integration of research and clinical practice.

Recently population of progenitor/stromal cells have been isolated form gingival connective tissue that shows stem cell nature and is known as Gingival Mesenchymal Stem Cells (GMSCs). GMSCs have shown to have higher rate of successive culture and proliferation compared to other sources of stem cells, and have demonstrated multi-lineage differentiation in osteoblastic, adipocytic, chondrocytic, endothelial and neural directions, however most of our present understanding and elucidation models stem from in vitro cell culture and in vivo animal models, which do not entirely translate to human clinical situations. To bridge our current knowledge gaps of tissue development processes, deeper understanding of biological processes is required, before reliable biologically based regenerative therapies become a clinical reality. Palatal gingival connective tissue, which can be a great source of GMSCs, is harvested primarily for treating gingival recession around teeth or dental implants. There is very little studied on the histological, cellular make up and the soft and hard tissue regenerative potential of this tissue owing to the presence of GMSCs. Also, the clinical decision as to where to harvest the tissue from relies on the amount of available tissue, indication of the treatment, and the clinical preference of the operator rather than based on progenitor potential and regenerative capabilities of the underlying cells.

Hence aim of this study is to investigate the progenitor potential of palatal GMSCs as well as characterizing and observing the functionality of isolated MSCs at two different palatal sites within the same patient.

The study will retrieve human soft tissue (gum tissue) samples from the roof of the mouth (palate) that are collected during soft tissue (gum) grafting surgical procedures routinely performed and are standard of care for treating gum recession in the School of Dentistry's Periodontology Clinic. For research purposes an additional 4mm of soft tissue samples will be obtained from two sites that is 2mm from front site (premolar) and 2mm from back site (molar) from the roof of the mouth (palate). The samples will be placed in sterile vials in the carrier medium and will be immediately transferred to the laboratory for the analysis. The remaining soft tissue (gum) graft will be used to cover the gum recession defects in that patient's mouth. A plastic guard will be placed on the roof of the mouth (palate) after the procedure to reduce post-op discomfort.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Patients needing soft tissue graft with teeth that have miller class I or II recession (>=2mm) on the facial aspects
* No previous harvesting procedure involving the palate
* Presence of periodontally healthy teeth at the recipient site.
* Ability of the participants to maintain good oral hygiene
* Patient not pregnant or breastfeeding
* Not taking medications known to cause gingival enlargement

Exclusion Criteria:

* Non-English speaking
* Smokers/tobacco users
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Patients that have severe gingival recession (Miller class III and IV) or < 2 mm.
* Previous harvesting procedure involving the palate (within 1 year)
* Presence of periodontal disease at the recipient site.
* Poor oral hygiene
* Patient pregnant or breastfeeding
* Taking medications known to cause gingival enlargement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Osteogenic potential | At day 1 Visit 1
  To assess mineralization (osteogenic) potential of mesenchymal stem cells isolated from premolar and molar site, double staining with alcian blue and von Kossa will be performed

SECONDARY OUTCOMES:
Adipogenic potential | At day 1 Visit 1
  To assess the adipogenic potential of mesenchymal stem cells isolated from premolar and molar site, cells will be stained with oil red o stain and the stained fat droplets will be visualized by light microscopy and photographed.
Genotype assay | At day 1 Visit 1
  RNA (ribonucleic acid) isolation and reverse transcriptase PCR (polymerase chain reaction) analysis will be performed to test the genetic make up of the mesenchymal stem cells isolated from premolar and molar site.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB School of Dentistry Department of Periodontology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No